CLINICAL TRIAL: NCT06199050
Title: The Effect of 360° Virtual Reality Movies on Fear and Anxiety
Acronym: ENGAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ENGAGE
Record Dates: First submitted 2023-06-16; First posted 2024-01-10 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Fear; Anxiety; Breast Cancer; Lung Cancer; Prostate Cancer; Head and Neck Cancer; Brain Tumor
MeSH Terms: conditions — Anxiety Disorders; Breast Neoplasms; Lung Neoplasms; Prostatic Neoplasms; Head and Neck Neoplasms; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 360° Virtual Reality Movies (Experimental): assess the amount of fear, anxiety and stress by using specific questionnaires:
  * SPecifIc RadIation Treatment related questions (SPIRIT)
  * Hospital Anxiety and Depression Scale (HADS)
  * Dutch version of the Questionnaire on stress symptoms (QSC-R23)
  General questions:
  * Education level
  * Marietal status
  * Medication use (in order to assess influence on fear)
  * Previous cancer diagnosis
  * Acquired information on treatment
  * Expected fear and anxiety mitigation strategies
  * Other cancer treatments (e.g. chemotherapy no, prior to RT, during RT, or after RT; surgery prior to or after RT)
  * PROM at baseline
  Clinical data:
  * Age
  * Gender
  * Cancer type
  * WHO status
  * TNM
  Interventions: Other: Questionnaire: SPIRIT; Other: Questionnaire: HADS; Other: Questionnaire: QSC-R23; Other: General questions; Other: Clinical data collected
- Group without intervention (Experimental): In a measurement over 5 months without any intervention the investigators have assessed the amount of fear, anxiety and stress by using a specific subjective questionnaire on the items below: assess the amount of fear, anxiety and stress by using specific questionnaires:
  * SPecifIc RadIation Treatment related questions (SPIRIT)
  * Hospital Anxiety and Depression Scale (HADS)
  * Dutch version of the Questionnaire on stress symptoms (QSC-R23)
  General questions:
  * Education level
  * Marietal status
  * Medication use (in order to assess influence on fear)
  * Previous cancer diagnosis
  * Acquired information on treatment
  * Expected fear and anxiety mitigation strategies
  * Other cancer treatments (e.g. chemotherapy no, prior to RT, during RT, or after RT; surgery prior to or after RT)
  * PROM at baseline
  Clinical data:
  * Age
  * Gender
  * Cancer type
  * WHO status
  * TNM
  Interventions: Other: Questionnaire: SPIRIT; Other: Questionnaire: HADS; Other: Questionnaire: QSC-R23; Other: General questions; Other: Clinical data collected

INTERVENTIONS:
Other: Questionnaire: SPIRIT — T0: Before the first intake at Maastro, the Trialpoli (TP) contacts a patient via phone to inform whether or not he is interested in participating in this study. If the patient shows interest in participating in the study, he will be invited for a consultation with the Trialpoli. This consultation takes place on the day of intake at Maastro. After consent, the patient is randomized to fill out T0 before or after the intake.
  T1: After filling out T0, the patient receives the ENGAGE information card with the url en QR code to the VR-movie. After watching the VR movie and before start RT the patient is asked to fill in T1. This questionnaire is distributed with instructions by the TP.
  T2: Between the 5th and the 15th radiation treatment, patients will be asked to fill in the questionnaires for the third and last time. The Patient Information Form (PIF) and Informed Consent (IC) are added in a separate document.
Other: Questionnaire: HADS — Hospital Anxiety and Depression Scale, 14 questions likert scale
Other: Questionnaire: QSC-R23 — Dutch version of the Questionnaire on stress symptoms, 23 questions likert scale
Other: General questions — * Education level
  * Marietal status
  * Medication use (in order to assess influence on fear)
  * Previous cancer diagnosis
  * Acquired information on treatment
  * Expected fear and anxiety mitigation strategies
  * Other cancer treatments (e.g. chemotherapy no, prior to RT, during RT, or after RT; surgery prior to or after RT)
  * PROM at baseline
Other: Clinical data collected — Clinical data in HIX:
  * Age
  * Gender
  * Cancer type
  * WHO status
  * TNM

SUMMARY:
To assess the effect of web-based 360° Virtual Reality movies on fear and anxiety, The investigators would like to assess the patient-perceived level of fear and anxiety quantitatively, making use of several questionnaires.

DETAILED DESCRIPTION:
In ENGAGE, a KWF Samenloop Voor Hoop subsidized project, we have developed VR movies to reduce fear and anxiety for patients who are going to be treated at Maastro. These movies are based on where most fear and anxiety are experienced and have been developed after extensive discussion with different disciplines in patient care and with agreement of the Director Patient Care. The movies include: 1) Mouldroom, 2) VMDIBH mamma photons, 3) Head and Neck photons, 4) Lung photons, 5) CT-scan, 6) Prostate photons, and 7) Head and Neck/ Neuro protons. Currently, the web-based 360° movies are implemented in clinical practice and the VR glasses with the 360° movies will be used as soon as social work has decided on where to integrate the use in the care pathway.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with breast- (only VMDIP), lung-, prostate-, head and neck cancer, a brain tumor.
* Age 18+
* Being able to speak, read and write in Dutch
* General interview between radiation oncologist and patient (= Intake)
* Ability to give written informed consent before the start of the study
* Decision talk about start of treatment must have taken place

Exclusion Criteria:

* Patients who are already receiving radiotherapy treatment
* Pre-operative consultation for breast cancer patients
* Patients who have seen the VR-videos already

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2025-05-13 (Actual); Study Completion 2025-05-13 (Actual)

PRIMARY OUTCOMES:
Subjective fear, anxiety and stress (QSC-R23) | 1 month
  What is the subjective fear, anxiety, and stress experience of patients before radiation treatment, specifically for the eight different user cases for which VR-movies are present, using the Questionnaire on Stress in Cancer Patients revised version (QSC-R23). Dutch version of the Questionnaire on stress symptoms (QSC-R23) - 23 questions likert scale.
Subjective fear, anxiety and stress (PROMS) | 1 month
  What is the subjective fear, anxiety, and stress experience of patients before radiation treatment, specifically for the eight different user cases for which VR-movies are present, using the Patient Reported Outcome Measures (PROMS) questionnaires. Patient reported outcome measures.
Subjective fear, anxiety and stress (HADS) | 1 month
  What is the subjective fear, anxiety, and stress experience of patients before radiation treatment, specifically for the eight different user cases for which VR-movies are present, using the Hospital Anxiety and Depression Scale (HADS). Hospital Anxiety and Depression Scale (HADS) - 14 questions likert scale
Subjective fear, anxiety and stress (SPIRIT) | 1 month
  What is the subjective fear, anxiety, and stress experience of patients before radiation treatment, specifically for the eight different user cases for which VR-movies are present, using the additional treatment-specific questions (SPIRIT). SPecifIc RadIation Treatment related questions (SPIRIT) - 10 questions likert scale
Relationship with demographics | 1 month
  Is there a relationship between fear, anxiety, stress experience, and the demographics of a patient.(I.e., prognosis, cancer indication, kind of treatment procedure)
Relationship between fear, anxiety, stress experience, and answers given in the standard PROMS questionnaire | 1 month
  Is there a relationship between fear, anxiety, stress experience, and answers given to specific questions in the standard PROMS questionnaire. (e.g., the general quality of life questionnaire (EQ5D), especially on FEAR and DEPRESSION and health-related quality of life (SF-36)?)

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Roumen, Study Director — Maastricht University; Maria Jacobs, Principal Investigator — Maastro
Locations (1):
- Maastricht Radiation Oncology, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided